CLINICAL TRIAL: NCT03787797
Title: Epicardial Adipose Tissue Thickness PredIcts Obstructive Coronary Artery Disease in Acute Coronary Syndrome Patients
Acronym: EPIC-ACS
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Amir Abbas Mahabadi, Principal Investigator, University Hospital, Essen
Other Study IDs: 18-8402-BO
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Epicardial adipose tissue; Chest pain; Echocardiography; Coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Coronary Artery Disease | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Assessment of epicardial adipose tissue thickness

SUMMARY:
Epicardial adipose tissue (EAT) is a visceral adipose tissue that surrounds the heart and the coronary arteries. It is metabolically active, secreting pro- and anti-inflammatory mediators and cytokines. With increasing EAT volume, inflammatory activity increasing, which suggests that EAT may locally influence atherosclerosis development in the coronary artery tree. The amount of EAT is associated with cardiovascular disease risk factors as well as presence and progression of subclinical atherosclerosis. Likewise, EAT volume is increased in patient with prevalent and incident coronary artery disease manifestation. In the setting of acute coronary syndrome, EAT was found to be associated with the TIMI risk score and Syntax II score. While CT imaging of the heart is the gold standard for EAT quantification, transthoracic echocardiography allows for a quick and reliable assessment of EAT thickness, as has been used in research studies and may qualify for routine EAT assessment in clinical routine.However, currently data on how quantification of EAT in clinical routine may impact patient management is lacking. We aim to investigate, whether quantification of EAT thickness via transthoracic echocardiography enables improved risk stratification in patients presenting with acute chest pain to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* admission to the emergency department of the University Hospital Essen with acute chest pain suggestive of an acute coronary syndrome

Exclusion Criteria:

* Known obstructive coronary artery disease prior to presentation, prior revascularization therapy, unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of patients without known coronary artery disease undergoing workup for suspected acute coronary syndrome at the emergency department of the University Hospital Essen.
Sampling Method: Probability Sample
Enrollment: 657 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Coronary revascularization | within 90 days after initial presentation
  Number of Participants with need for coronary revascularization therapy

SECONDARY OUTCOMES:
Invasive coronary angiography | within 90 days after initial presentation
  Number of Participants undergoing invasive coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Amir A Mahabadi, MD, Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available upon request.

REFERENCES:
- [Derived] Roggel A, Jehn S, Dykun I, Balcer B, Al-Rashid F, Totzeck M, Risse J, Kill C, Rassaf T, Mahabadi A. Regional wall motion abnormalities on focused transthoracic echocardiography in patients presenting with acute chest pain: a predefined post hoc analysis of the prospective single-centre observational EPIC-ACS study. BMJ Open. 2024 Sep 10;14(9):e085677. doi: 10.1136/bmjopen-2024-085677. PMID 39260858